CLINICAL TRIAL: NCT03014336
Title: A New and Innovative Method for CO2 Removal in Anesthetic Circuits:
Brief Title: A New and Innovative Method for CO2 Removal in Anesthetic Circuits: Replacing Chemical Granulate
Acronym: memsorb
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: DMF Medical Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DMF-CLIN-16-01
Record Dates: First submitted 2016-10-12; First posted 2017-01-09 (Estimated); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Anesthesia
Keywords: co2 removal, anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Patients receive standard care with a standard CO2 absorber and agree to include their data in the study.
- memsorb (Experimental): Patients agree to receive standard care but using memsorb, the new CO2 filter evaluated in this study.
  Interventions: Device: memsorb

INTERVENTIONS:
Device: memsorb — memsorb is a CO2 filter replacing current chemical CO2 absorbers
  Arms: memsorb

SUMMARY:
The drawbacks of chemical CO2 absorbers include the production of compounds harmful to patients that also lead into increased cost and environmental impact, as well as the daily disposal of compound special waste. Sustainable management of general anesthesia is a growing concern. Continually diluting anesthetic circuits, and the disposal of chemical granulate are serious environmental problems.

DETAILED DESCRIPTION:
DMF Medical has developed a next-generation CO2 filter in order to address the safety issues with current chemical CO2 absorbers in anesthesia.

memsorb uses patented advanced medical membrane technology to filter CO2 from anesthetic circuits rather than absorbing via a chemical reaction.

This game changing technology relies on a polymeric membrane core (similar to the ones used in oxygenators for cardiac surgery) that selectively allows CO2 to leave the rebreathing system, while maintaining the anesthetic vapor in the circuit.

memsorb is a cartridge similar in size and shape to current solutions that simply clicks in place.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Physical Status Class I, II, III (low-medium risk patient)
* English-speaking patients

Exclusion Criteria:

* Self-reported as pregnant
* American Society of Anesthesiologists Physical Status Class IV (high risk patient)
* Patients scheduled for emergency surgery
* Documented respiratory disease, including COPD and severe asthma
* Documented elevated pressure in the brain (intra cranial pressure, ICP)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2017-01; Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
End Tidal CO2 | Up to 12h
  Concentration of carbon dioxide during expiratory cycle.

OTHER OUTCOMES:
Fresh gas flow | Up to 12h
  Analysis of fresh gas flow into the machine.
Fractional concentration of inspired CO2 | Up to 12h
  Analysis of concentration of CO2 during inspiratory cycle.
Fractional concentration of inspired O2 | Up to 12h
  Analysis of concentration of O2 in inspired gas.
Arterial blood oxygen saturation | Up to 12h
  Saturation of oxygen in arterial blood where measured by pulse oximetry and/or blood gas analysis.
Arterial blood CO2 partial pressure | Up to 12h
  Saturation of carbon dioxide in arterial blood measured by a blood gas analyzer.
pH measurement | Single collected measurement not more than 60 min after extubation
  pH of the condensed water in the drain valve and the PAL filter.
Length of surgery | Up to 12h
  Duration of surgical procedure.
Ventilation frequency | Up to 12h
  Measurement of patient breathing rate.
Ventilation pressure | Up to 12h
  Measurement of patient inspiratory pressure.
Tidal volume | Up to 12h
  Measurement of total lung volume as represented by the volume of air displaced between normal inhalation and exhalation.
Patient temperature | Up to 12h
  Body temperature of patient.
Relaxation status | Up to 12h
  Neuromuscular relaxation of patient.
Heart rate | Up to 12h
  Measurement and collection of patient heart rate.
Blood pressure | Up to 12h
  Measurement and collection of patient mean, systolic and diastolic blood pressure.
Patient weight | during preoperative assessment
  Weight of patient as collected from anaesthesia patient record database.
Patient height | during preoperative assessment
  Height of patient as collected from anaesthesia patient record database.
Patient age | during preoperative assessment
  Age of patient as collected from anaesthesia patient record database.
Patient medications | during preoperative assessment
  Medications being taken by patient as collected from anaesthesia patient record database.
Lung disease | during preoperative assessment
  Incidence of lung disease as collected from anaesthesia patient record database.
Anaesthetic agent | Up to 12h
  Inhaled and exhaled fraction of anaesthetic agent as collected from the anaesthetic patient record database

CONTACTS AND LOCATIONS:
Overall Officials: Orlando Hung, MD, Principal Investigator — Nova Scotia Health Authority
Locations (2):
- Canada (2):
  - Queen Elizabeth II HSC, Halifax Infirmary Site, Halifax, Nova Scotia
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No